CLINICAL TRIAL: NCT04765813
Title: A Randomized Clinical Trial to Assess the Efficacy of a Psychological Treatment to Quit Smoking Assisted With an App
Brief Title: Use of a Smartphone Application (App) to Assist a Cognitive-Behavioral Smoking Cessation Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Principal Investigator, Elisardo Becoña Iglesias, Professor of Clinical Psychology at the Faculty of Psychology, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PID2019-109400RB-I00
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT and active smartphone mobile application (Experimental): Participants receive a cognitive-behavioral treatment to quit smoking along with an App with active therapeutic components
  Interventions: Behavioral: Cognitive-behavioral treatment to quit smoking along with an App with active therapeutic components
- CBT and control smartphone mobile application (Active Comparator): Participants receive a cognitive-behavioral treatment to quit smoking along with a control App
  Interventions: Behavioral: Cognitive-behavioral treatment to quit smoking along with a control App

INTERVENTIONS:
Behavioral: Cognitive-behavioral treatment to quit smoking along with an App with active therapeutic components — Cognitive-behavioral smoking cessation treatment components will be: treatment contract, self-report and graphic representation of cigarette consumption, information about tobacco, stimulus control, activities for the avoidance of withdrawal syndrome, physiological feedback (CO in expired air) on cigarette consumption, nicotine fading (change of cigarette brands each week progressively decreasing the intake of nicotine and tar), and relapse-prevention strategies (assertion training, problem-solving training, change tobacco-related misconceptions, management of anxiety and anger, exercise, weight control, self-reinforcing, and changing irrational beliefs).
  Participants will use a smartphone App with therapeutic components during the intervention (8 weeks) and follow-up period (time frame: one year).
  Arms: CBT and active smartphone mobile application
Behavioral: Cognitive-behavioral treatment to quit smoking along with a control App — Cognitive-behavioral smoking cessation treatment components will be: treatment contract, self-report and graphic representation of cigarette consumption, information about tobacco, stimulus control, activities for the avoidance of withdrawal syndrome, physiological feedback (CO in expired air) on cigarette consumption, nicotine fading (change of cigarette brands each week progressively decreasing the intake of nicotine and tar), and relapse-prevention strategies (assertion training, problem-solving training, change tobacco-related misconceptions, management of anxiety and anger, exercise, weight control, self-reinforcing, and changing irrational beliefs).
  Participants will use a control smartphone App (only to access session materials) during the intervention period (8 weeks).
  Arms: CBT and control smartphone mobile application

SUMMARY:
This randomized controlled clinical trial examines the effectiveness of a face-to-face* cognitive-behavioral behavioral treatment to quit smoking enriched with an App. This project aims to innovate in the psychological smoking cessation treatment and increase abstinence rates in the short and long term.

* Due to the COVID-19 the face-to-face treatment will be conducted in an online format.

DETAILED DESCRIPTION:
Psychological treatment (cognitive-behavioral) is a first-line smoking cessation treatment that has proven its efficacy. However, it is necessary to continue investigating to improve smoking outcomes as abstinence and reduce relapse rates. The use of information technologies (ICTs) in the field of health has grown and developed significantly in recent years. Specifically, mobile applications (Apps), aimed at different health-related aspects (mHealth Apps), are a valuable resource. Its use, as a complement to the face-to-face treatment, could help to increase motivation to quit smoking, treatment adherence, and therapeutic activities compliance.

mHealth Apps are becoming highly relevant due to their cost-effectiveness and the added attractiveness for many users. Considering this context, the main aim of the present project is to design and assess the efficacy of a cognitive-behavioral treatment (CBT) for smoking cessation enriched with a Smartphone App.

A randomized clinical trial will be carried out with a sample of 270 treatment-seeking smokers at the Smoking Cessation and Addictive Disorders Unit of the University of Santiago de Compostela. Participants will be randomly assigned to one of the following groups:

1. The experimental group (CBT + App), in which participants will receive a cognitive-behavioral treatment* to quit smoking along with an App with active therapeutic components during the treatment and 12 months follow-ups period (n = 135)
2. The control group (CBT), in which participants will receive the same cognitive-behavioral treatment* along with the use of a Control App (without active components) during the treatment (n = 135).

The main hypothesis is that the combination of a cognitive-behavioral psychological treatment to quit smoking and an App with active therapeutic components will obtain higher abstinence rates at the end of treatment and the 12-month follow-up period, compared to the control group

* Due to the COVID-19, the face-to-face cognitive-behavioral treatment will be conducted in an online format

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older who smoke at least 8 cigarettes per day
* Desire to participate voluntarily in the treatment offered to quit smoking
* Correctly fill out all the pretreatment assessment questionnaires
* Be able to provide written informed consent
* Currently own a valid email and a smartphone Android or iOS and willing to use it during treatment

Exclusion Criteria:

* To have a diagnosis of a severe mental disorder (bipolar disorder and/or psychotic disorder)
* To have a substance use disorder (alcohol, cannabis, cocaine, heroin), different from a tobacco use disorder
* To smoke rolling snuff, cigars, little cigars, or other tobacco products
* To have participated in an effective psychological treatment to quit smoking during the previous 12 months
* To have received other effective pharmacological treatment to quit smoking in the previous 12 months (nicotine gum or patches, bupropion, varenicline)
* To have a physical pathology involving life-threatening risks for the person who would require immediate intervention in individual format (e.g., recent myocardial infarction, pneumothorax)
* To have a visual impairment that impedes the use of the App

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Point-prevalence abstinence | 1 year
  Participants will be considered abstinent if they report abstinence, not even a puff of a cigarette, for ≥7 days at the end of treatment (week 8 since beginning treatment), and prior to follow-up day at 3-, 6-, and 12-months follow-up.

SECONDARY OUTCOMES:
Continuous abstinence | 1 year
  Self-reported 30-day point prevalence abstinence at 3-, 6-, and 12-month follow-up
Reduction of cigarette consumption (cigarettes per day) | 1 year
  Reduction of cigarette consumption between baseline and each follow-up will be calculated from the number of cigarettes smoked in the past 7 days at the end of treatment (week 8 since beginning treatment) and at 3-, 6-, and 12-months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Elisardo Becoña, PhD, Principal Investigator — University of Santiago de Compostela
Locations (1):
- Smoking Cessation and Addictive Disorders Unit, Faculty of Psychology, University of Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopez-Duran A, Becona E, Senra C, Suarez-Castro D, Barroso-Hurtado M, Martinez-Vispo C. A Randomized Clinical Trial to Assess the Efficacy of a Psychological Treatment to Quit Smoking Assisted with an App: Study Protocol. Int J Environ Res Public Health. 2022 Aug 8;19(15):9770. doi: 10.3390/ijerph19159770. PMID 35955123
- [Derived] Lopez-Duran A, Martinez-Vispo C, Barroso-Hurtado M, Suarez-Castro D, Becona E. Incorporating technology in smoking cessation interventions: In-person vs. Video-call formats. Int J Med Inform. 2025 Mar;195:105774. doi: 10.1016/j.ijmedinf.2024.105774. Epub 2024 Dec 24. PMID 39742855